CLINICAL TRIAL: NCT01777542
Title: Pharmacological Treatment of Rett Syndrome by Stimulation of Synaptic Maturation With Recombinant Human IGF-1(Mecasermin [rDNA] Injection)
Brief Title: Treatment of Rett Syndrome With Recombinant Human IGF-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: International Rett Syndrome Foundation (Other)
Responsible Party: Principal Investigator, Mustafa Sahin, Associate Professor of Neurology, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-P00005610
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; RTT; IGF-1; autism spectrum disorder
MeSH Terms: conditions — Rett Syndrome; Autism Spectrum Disorder | interventions — mecasermin; DNA, Ribosomal; Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Period 1 (Active Comparator): One half of subjects will be randomly assigned to receive Recombinant Human Insulin Growth Factor 1 (rhIGF-1) , and the other half of subjects will be randomly assigned to receive placebo.
  Interventions: Drug: Recombinant Human Insulin Growth Factor 1 (rhIGF-1); Drug: Placebo
- Treatment Period 2 (Placebo Comparator): Subjects that initially received Recombinant Human Insulin Growth Factor 1 (rhIGF-1) will now receive placebo, and subjects that initially received placebo will now receive Recombinant Human Insulin Growth Factor 1 (rhIGF-1).
  Interventions: Drug: Recombinant Human Insulin Growth Factor 1 (rhIGF-1); Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Human Insulin Growth Factor 1 (rhIGF-1) — Subjects will receive twice daily subcutaneous injections of IGF-1.
  Other Names: mecasermin [rDNA] injection; Increlex
Drug: Placebo — Subjects will receive twice daily subcutaneous injections of a saline solution (placebo).
  Other Names: saline

SUMMARY:
Investigators are recruiting children for a clinical trial using the medication recombinant human IGF-1 (a.k.a. mecasermin or INCRELEX) to see if it improves the health of children with Rett syndrome (RTT). While IGF-1 is approved by the Food & Drug Administration (FDA) for certain use in children, it is considered an investigational drug in this trial because it has not previously been used to treat RTT. Information from this study will help determine if IGF-1 effectively treats RTT but will not necessarily lead to FDA approval of IGF-1 as a treatment for RTT.

DETAILED DESCRIPTION:
Enrolled subjects will complete five study periods: screening, two 20-week long treatment periods, a 28-week break between treatment periods ("washout"), and a follow-up phone call 4 weeks after all treatment ends. Subjects will be chosen at random to receive either IGF-1 or placebo during the first treatment period and then switch to the alternate medication for the second treatment period. Therefore, by completion of the trial, all subjects will have received treatment with IGF-1 for 20 weeks. The study will be double-blinded; meaning, neither subjects' families nor study investigators will know who is receiving IGF-1 or placebo at any time. Treatment must be administered by the caregiver twice daily through subcutaneous (just underneath the skin) injections. Caregivers will be trained by research nurses in how to administer the medication. Participation in this study will last approximately eighteen months.

Throughout the course of the trial, investigators will collect information to assess the effects of IGF-1 and monitor for safety. Families must attend study visits at Boston Children's Hospital a total of seven times (including the screening visit) over the course of 18 months. These visits cannot be completed at any other hospital. Parents will fill out questionnaires and undergo a structured interview reporting on their child's health, behavior, and mood. Subjects will undergo clinical and physical examinations by a study doctor. Non-invasive devices and cameras will also be used to monitor things like breathing, hand movements, heart rate, and body temperature. Blood and urine will be collected for routine laboratory tests to monitor for safety. Investigators will also monitor safety by asking parents to complete a medication diary and side effect reporting form on a regular basis. Between trips to Boston Children's Hospital, parents will complete a set of online questionnaires and undergo a structured interview over the phone.

The cost of travel and lodging during research-related visits to and from the hospital will not be covered by the study. If a condition or illness is identified during the trial (and is determined to be unrelated to study treatments), referrals to outside medical care will be made. Study medications and all research-related materials and services will be provided at no cost to participants. Parking vouchers will be provided for all study-related hospital visits.

The study is investigating 5 potential effects:

1. IGF-1 may improve subjects' behavior, communication and/or mood. In order to measure this, investigators will evaluate subjects every 5 weeks throughout each treatment period with behavioral and psychological assessments. All of the tests used during these evaluations are non-invasive. Investigators will ask parents what their impressions are about their child's behavior and day-to-day activities through a structured parental interview and various questionnaires.
2. Investigators will examine subjects' brain function through use of a brain- monitoring device known as electroencephalography (EEG). The EEG measurements will be taken while investigators present subjects with exercises to stimulate their vision and hearing. EEG is a non-invasive way of recording the electrical activity of a subject's brain by applying a net of monitors (electrodes) to their scalp. Through this method investigators gain insight into how brain processes visual and auditory stimulus.
3. As one of the features of RTT is unstable vital signs, investigators are trying to determine if IGF-1 has any effect on normalizing subjects' heart rate and breathing patterns. To measure this, investigators will ask subjects to wear a non-invasive device that includes three electrocardiogram connectors and two stretchy bands that wrap around her chest and abdomen to measure heart rate and respiratory patterns.
4. The safety of IGF-1 in children with RTT is very important. Investigators will ask parents to complete a medication diary and side effect reporting form on a regular basis. In addition, laboratory tests will be performed every 10 weeks throughout each treatment period to evaluate the safety of IGF-1. These will be blood tests similar to those provided in typical clinical care. Subjects will undergo regular non-invasive comprehensive physical and neurological examinations, tonsil evaluation, electrocardiogram (ECG), echocardiogram, scoliosis x-ray, bone age x-ray, ophthalmological exam, and measurements of height, weight and head circumference.
5. Children with RTT often experience unintended, stereotyped hand movements. The Qsensor® is a non-invasive device worn on a fabric bracelet that continually measures subjects' movement. Investigators will use the Qsensor® to determine whether or not IGF-1 affects the presentation of stereotyped hand movements. As such, investigators will ask subjects to wear the Qsensor® during study visits every 10 weeks throughout each treatment period and occasionally at home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "classic" (or "typical") Rett Syndrome
* Genetic documentation of MECP2 mutation
* Subject must be post-regression (Hagberg Stage 2)
* Subject and caregiver's primary language must be English
* Subject must reside in North America (US and Canada)
* Caregiver must have internet access and be able to complete questionnaires online and communicate via email
* Subject is stable on current medications for at least 4 weeks
* Subject's regimen of non-pharmacological interventions (physical therapy, speech therapy, etc.) is stable for at least 90 days

Exclusion Criteria:

* Severe scoliosis (curvature >40 degrees)
* Bone-age greater than 11 years
* Cardiomegaly (enlarged heart)
* Tanner stage 2 or higher breast development
* Allergy to IGF-1
* Prior use of IGF-1, growth hormone, or sex steroids

Ages: 2 Years to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sahin, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Khwaja OS, Ho E, Barnes KV, O'Leary HM, Pereira LM, Finkelstein Y, Nelson CA 3rd, Vogel-Farley V, DeGregorio G, Holm IA, Khatwa U, Kapur K, Alexander ME, Finnegan DM, Cantwell NG, Walco AC, Rappaport L, Gregas M, Fichorova RN, Shannon MW, Sur M, Kaufmann WE. Safety, pharmacokinetics, and preliminary assessment of efficacy of mecasermin (recombinant human IGF-1) for the treatment of Rett syndrome. Proc Natl Acad Sci U S A. 2014 Mar 25;111(12):4596-601. doi: 10.1073/pnas.1311141111. Epub 2014 Mar 12. PMID 24623853
- [Background] Schultz RJ, Glaze DG, Motil KJ, Armstrong DD, del Junco DJ, Hubbard CR, Percy AK. The pattern of growth failure in Rett syndrome. Am J Dis Child. 1993 Jun;147(6):633-7. doi: 10.1001/archpedi.1993.02160300039018. PMID 8506830
- [Background] Williamson SL, Christodoulou J. Rett syndrome: new clinical and molecular insights. Eur J Hum Genet. 2006 Aug;14(8):896-903. doi: 10.1038/sj.ejhg.5201580. PMID 16865103
- [Background] Weese-Mayer DE, Lieske SP, Boothby CM, Kenny AS, Bennett HL, Silvestri JM, Ramirez JM. Autonomic nervous system dysregulation: breathing and heart rate perturbation during wakefulness in young girls with Rett syndrome. Pediatr Res. 2006 Oct;60(4):443-9. doi: 10.1203/01.pdr.0000238302.84552.d0. Epub 2006 Aug 28. PMID 16940240
- [Background] Percy AK. Clinical trials and treatment prospects. Ment Retard Dev Disabil Res Rev. 2002;8(2):106-11. doi: 10.1002/mrdd.10022. PMID 12112736
- [Background] Amir RE, Van den Veyver IB, Wan M, Tran CQ, Francke U, Zoghbi HY. Rett syndrome is caused by mutations in X-linked MECP2, encoding methyl-CpG-binding protein 2. Nat Genet. 1999 Oct;23(2):185-8. doi: 10.1038/13810. PMID 10508514
- [Background] Nan X, Ng HH, Johnson CA, Laherty CD, Turner BM, Eisenman RN, Bird A. Transcriptional repression by the methyl-CpG-binding protein MeCP2 involves a histone deacetylase complex. Nature. 1998 May 28;393(6683):386-9. doi: 10.1038/30764. PMID 9620804
- [Background] Shahbazian MD, Antalffy B, Armstrong DL, Zoghbi HY. Insight into Rett syndrome: MeCP2 levels display tissue- and cell-specific differences and correlate with neuronal maturation. Hum Mol Genet. 2002 Jan 15;11(2):115-24. doi: 10.1093/hmg/11.2.115. PMID 11809720
- [Background] Cohen DR, Matarazzo V, Palmer AM, Tu Y, Jeon OH, Pevsner J, Ronnett GV. Expression of MeCP2 in olfactory receptor neurons is developmentally regulated and occurs before synaptogenesis. Mol Cell Neurosci. 2003 Apr;22(4):417-29. doi: 10.1016/s1044-7431(03)00026-5. PMID 12727440
- [Background] Gemelli T, Berton O, Nelson ED, Perrotti LI, Jaenisch R, Monteggia LM. Postnatal loss of methyl-CpG binding protein 2 in the forebrain is sufficient to mediate behavioral aspects of Rett syndrome in mice. Biol Psychiatry. 2006 Mar 1;59(5):468-76. doi: 10.1016/j.biopsych.2005.07.025. Epub 2005 Sep 30. PMID 16199017
- [Background] Guy J, Hendrich B, Holmes M, Martin JE, Bird A. A mouse Mecp2-null mutation causes neurological symptoms that mimic Rett syndrome. Nat Genet. 2001 Mar;27(3):322-6. doi: 10.1038/85899. PMID 11242117
- [Background] Shahbazian M, Young J, Yuva-Paylor L, Spencer C, Antalffy B, Noebels J, Armstrong D, Paylor R, Zoghbi H. Mice with truncated MeCP2 recapitulate many Rett syndrome features and display hyperacetylation of histone H3. Neuron. 2002 Jul 18;35(2):243-54. doi: 10.1016/s0896-6273(02)00768-7. PMID 12160743
- [Background] Giacometti E, Luikenhuis S, Beard C, Jaenisch R. Partial rescue of MeCP2 deficiency by postnatal activation of MeCP2. Proc Natl Acad Sci U S A. 2007 Feb 6;104(6):1931-6. doi: 10.1073/pnas.0610593104. Epub 2007 Jan 31. PMID 17267601
- [Background] Chao HT, Zoghbi HY, Rosenmund C. MeCP2 controls excitatory synaptic strength by regulating glutamatergic synapse number. Neuron. 2007 Oct 4;56(1):58-65. doi: 10.1016/j.neuron.2007.08.018. PMID 17920015
- [Background] Dani VS, Chang Q, Maffei A, Turrigiano GG, Jaenisch R, Nelson SB. Reduced cortical activity due to a shift in the balance between excitation and inhibition in a mouse model of Rett syndrome. Proc Natl Acad Sci U S A. 2005 Aug 30;102(35):12560-5. doi: 10.1073/pnas.0506071102. Epub 2005 Aug 22. PMID 16116096
- [Background] Nelson ED, Kavalali ET, Monteggia LM. MeCP2-dependent transcriptional repression regulates excitatory neurotransmission. Curr Biol. 2006 Apr 4;16(7):710-6. doi: 10.1016/j.cub.2006.02.062. PMID 16581518
- [Background] Chang Q, Khare G, Dani V, Nelson S, Jaenisch R. The disease progression of Mecp2 mutant mice is affected by the level of BDNF expression. Neuron. 2006 Feb 2;49(3):341-8. doi: 10.1016/j.neuron.2005.12.027. PMID 16446138
- [Background] Schuman EM. Neurotrophin regulation of synaptic transmission. Curr Opin Neurobiol. 1999 Feb;9(1):105-9. doi: 10.1016/s0959-4388(99)80013-0. PMID 10072368
- [Background] Bondy CA. Transient IGF-I gene expression during the maturation of functionally related central projection neurons. J Neurosci. 1991 Nov;11(11):3442-55. doi: 10.1523/JNEUROSCI.11-11-03442.1991. PMID 1658250
- [Background] Liu JP, Baker J, Perkins AS, Robertson EJ, Efstratiadis A. Mice carrying null mutations of the genes encoding insulin-like growth factor I (Igf-1) and type 1 IGF receptor (Igf1r). Cell. 1993 Oct 8;75(1):59-72. PMID 8402901
- [Background] Tropea D, Kreiman G, Lyckman A, Mukherjee S, Yu H, Horng S, Sur M. Gene expression changes and molecular pathways mediating activity-dependent plasticity in visual cortex. Nat Neurosci. 2006 May;9(5):660-8. doi: 10.1038/nn1689. Epub 2006 Apr 23. PMID 16633343
- [Background] Yoshii A, Constantine-Paton M. BDNF induces transport of PSD-95 to dendrites through PI3K-AKT signaling after NMDA receptor activation. Nat Neurosci. 2007 Jun;10(6):702-11. doi: 10.1038/nn1903. Epub 2007 May 21. PMID 17515902
- [Background] Zheng WH, Quirion R. Comparative signaling pathways of insulin-like growth factor-1 and brain-derived neurotrophic factor in hippocampal neurons and the role of the PI3 kinase pathway in cell survival. J Neurochem. 2004 May;89(4):844-52. doi: 10.1111/j.1471-4159.2004.02350.x. PMID 15140184
- [Background] Ramsey MM, Adams MM, Ariwodola OJ, Sonntag WE, Weiner JL. Functional characterization of des-IGF-1 action at excitatory synapses in the CA1 region of rat hippocampus. J Neurophysiol. 2005 Jul;94(1):247-54. doi: 10.1152/jn.00768.2004. PMID 15985695
- [Background] Xing C, Yin Y, Chang R, Gong X, He X, Xie Z. Effects of insulin-like growth factor 1 on synaptic excitability in cultured rat hippocampal neurons. Exp Neurol. 2007 May;205(1):222-9. doi: 10.1016/j.expneurol.2007.01.029. Epub 2007 Feb 7. PMID 17335809
- [Background] Riikonen R, Makkonen I, Vanhala R, Turpeinen U, Kuikka J, Kokki H. Cerebrospinal fluid insulin-like growth factors IGF-1 and IGF-2 in infantile autism. Dev Med Child Neurol. 2006 Sep;48(9):751-5. doi: 10.1017/S0012162206001605. PMID 16904022
- [Background] Acampa M, Guideri F. Cardiac disease and Rett syndrome. Arch Dis Child. 2006 May;91(5):440-3. doi: 10.1136/adc.2005.090290. PMID 16632674
- [Background] Johnston MV, Jeon OH, Pevsner J, Blue ME, Naidu S. Neurobiology of Rett syndrome: a genetic disorder of synapse development. Brain Dev. 2001 Dec;23 Suppl 1:S206-13. doi: 10.1016/s0387-7604(01)00351-5. PMID 11738874
- [Background] Kaufmann WE, Taylor CV, Hohmann CF, Sanwal IB, Naidu S. Abnormalities in neuronal maturation in Rett syndrome neocortex: preliminary molecular correlates. Eur Child Adolesc Psychiatry. 1997;6 Suppl 1:75-7. PMID 9452926
- [Background] Kaufmann WE, MacDonald SM, Altamura CR. Dendritic cytoskeletal protein expression in mental retardation: an immunohistochemical study of the neocortex in Rett syndrome. Cereb Cortex. 2000 Oct;10(10):992-1004. doi: 10.1093/cercor/10.10.992. PMID 11007550
- [Background] Tropea D, Giacometti E, Wilson NR, Beard C, McCurry C, Fu DD, Flannery R, Jaenisch R, Sur M. Partial reversal of Rett Syndrome-like symptoms in MeCP2 mutant mice. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):2029-34. doi: 10.1073/pnas.0812394106. PMID 19208815
- [Background] Julu PO, Kerr AM, Apartopoulos F, Al-Rawas S, Engerstrom IW, Engerstrom L, Jamal GA, Hansen S. Characterisation of breathing and associated central autonomic dysfunction in the Rett disorder. Arch Dis Child. 2001 Jul;85(1):29-37. doi: 10.1136/adc.85.1.29. PMID 11420195
- [Background] Chen RZ, Akbarian S, Tudor M, Jaenisch R. Deficiency of methyl-CpG binding protein-2 in CNS neurons results in a Rett-like phenotype in mice. Nat Genet. 2001 Mar;27(3):327-31. doi: 10.1038/85906. PMID 11242118
- [Background] Castro J, Garcia RI, Kwok S, Banerjee A, Petravicz J, Woodson J, Mellios N, Tropea D, Sur M. Functional recovery with recombinant human IGF1 treatment in a mouse model of Rett Syndrome. Proc Natl Acad Sci U S A. 2014 Jul 8;111(27):9941-6. doi: 10.1073/pnas.1311685111. Epub 2014 Jun 23. PMID 24958891
- [Background] Pini G, Scusa MF, Congiu L, Benincasa A, Morescalchi P, Bottiglioni I, Di Marco P, Borelli P, Bonuccelli U, Della-Chiesa A, Prina-Mello A, Tropea D. IGF1 as a Potential Treatment for Rett Syndrome: Safety Assessment in Six Rett Patients. Autism Res Treat. 2012;2012:679801. doi: 10.1155/2012/679801. Epub 2012 Jun 13. PMID 22934177
- [Background] Lopez-Lopez C, LeRoith D, Torres-Aleman I. Insulin-like growth factor I is required for vessel remodeling in the adult brain. Proc Natl Acad Sci U S A. 2004 Jun 29;101(26):9833-8. doi: 10.1073/pnas.0400337101. Epub 2004 Jun 21. PMID 15210967
- [Background] Aberg MA, Aberg ND, Hedbacker H, Oscarsson J, Eriksson PS. Peripheral infusion of IGF-I selectively induces neurogenesis in the adult rat hippocampus. J Neurosci. 2000 Apr 15;20(8):2896-903. doi: 10.1523/JNEUROSCI.20-08-02896.2000. PMID 10751442
- [Background] Pan W, Kastin AJ. Interactions of IGF-1 with the blood-brain barrier in vivo and in situ. Neuroendocrinology. 2000 Sep;72(3):171-8. doi: 10.1159/000054584. PMID 11025411
- [Background] Kaufmann WE, Tierney E, Rohde CA, Suarez-Pedraza MC, Clarke MA, Salorio CF, Bibat G, Bukelis I, Naram D, Lanham DC, Naidu S. Social impairments in Rett syndrome: characteristics and relationship with clinical severity. J Intellect Disabil Res. 2012 Mar;56(3):233-47. doi: 10.1111/j.1365-2788.2011.01404.x. Epub 2011 Mar 8. PMID 21385260
- [Background] Mount RH, Charman T, Hastings RP, Reilly S, Cass H. The Rett Syndrome Behaviour Questionnaire (RSBQ): refining the behavioural phenotype of Rett syndrome. J Child Psychol Psychiatry. 2002 Nov;43(8):1099-110. doi: 10.1111/1469-7610.00236. PMID 12455930
- [Background] Esbensen AJ, Rojahn J, Aman MG, Ruedrich S. Reliability and validity of an assessment instrument for anxiety, depression, and mood among individuals with mental retardation. J Autism Dev Disord. 2003 Dec;33(6):617-29. doi: 10.1023/b:jadd.0000005999.27178.55. PMID 14714931
- [Background] Rojahn J, Rowe EW, Kasdan S, Moore L, van Ingen DJ. Psychometric properties of the Aberrant Behavior Checklist, the Anxiety, Depression and Mood Scale, the Assessment of Dual Diagnosis and the Social Performance Survey Schedule in adults with intellectual disabilities. Res Dev Disabil. 2011 Nov-Dec;32(6):2309-20. doi: 10.1016/j.ridd.2011.07.035. Epub 2011 Sep 1. PMID 21889296
- [Background] Barnes KV, Coughlin FR, O'Leary HM, Bruck N, Bazin GA, Beinecke EB, Walco AC, Cantwell NG, Kaufmann WE. Anxiety-like behavior in Rett syndrome: characteristics and assessment by anxiety scales. J Neurodev Disord. 2015;7(1):30. doi: 10.1186/s11689-015-9127-4. Epub 2015 Sep 15. PMID 26379794
- [Background] Hagberg B. Clinical manifestations and stages of Rett syndrome. Ment Retard Dev Disabil Res Rev. 2002;8(2):61-5. doi: 10.1002/mrdd.10020. PMID 12112728
- [Background] McCracken JT, McGough J, Shah B, Cronin P, Hong D, Aman MG, Arnold LE, Lindsay R, Nash P, Hollway J, McDougle CJ, Posey D, Swiezy N, Kohn A, Scahill L, Martin A, Koenig K, Volkmar F, Carroll D, Lancor A, Tierney E, Ghuman J, Gonzalez NM, Grados M, Vitiello B, Ritz L, Davies M, Robinson J, McMahon D; Research Units on Pediatric Psychopharmacology Autism Network. Risperidone in children with autism and serious behavioral problems. N Engl J Med. 2002 Aug 1;347(5):314-21. doi: 10.1056/NEJMoa013171. PMID 12151468
- [Background] Arnold LE, Vitiello B, McDougle C, Scahill L, Shah B, Gonzalez NM, Chuang S, Davies M, Hollway J, Aman MG, Cronin P, Koenig K, Kohn AE, McMahon DJ, Tierney E. Parent-defined target symptoms respond to risperidone in RUPP autism study: customer approach to clinical trials. J Am Acad Child Adolesc Psychiatry. 2003 Dec;42(12):1443-50. doi: 10.1097/00004583-200312000-00011. PMID 14627879
- [Background] Arnold LE, Wender PH, McCloskey K, Snyder SH. Levoamphetamine and dextroamphetamine: comparative efficacy in the hyperkinetic syndrome. Assessment by target symptoms. Arch Gen Psychiatry. 1972 Dec;27(6):816-22. doi: 10.1001/archpsyc.1972.01750300078015. No abstract available. PMID 4564954
- [Background] Arnold LE, Christopher J, Huestis R, Smeltzer DJ. Methylphenidate vs dextroamphetamine vs caffeine in minimal brain dysfunction: controlled comparison by placebo washout design with Bayes' analysis. Arch Gen Psychiatry. 1978 Apr;35(4):463-73. doi: 10.1001/archpsyc.1978.01770280073008. PMID 365123
- [Background] Arnold LE, Huestis RD, Smeltzer DJ, Scheib J, Wemmer D, Colner G. Levoamphetamine vs dextroamphetamine in minimal brain dysfunction. Replication, time response, and differential effect by diagnostic group and family rating. Arch Gen Psychiatry. 1976 Mar;33(3):292-301. doi: 10.1001/archpsyc.1976.01770030012002. PMID 769721
- [Background] Bebbington A, Anderson A, Ravine D, Fyfe S, Pineda M, de Klerk N, Ben-Zeev B, Yatawara N, Percy A, Kaufmann WE, Leonard H. Investigating genotype-phenotype relationships in Rett syndrome using an international data set. Neurology. 2008 Mar 11;70(11):868-75. doi: 10.1212/01.wnl.0000304752.50773.ec. PMID 18332345
- [Background] Fidler DJ, Hepburn S, Rogers S. Early learning and adaptive behaviour in toddlers with Down syndrome: evidence for an emerging behavioural phenotype? Downs Syndr Res Pract. 2006 Jun;9(3):37-44. doi: 10.3104/reports.297. PMID 16869373
- [Background] Mirrett PL, Bailey DB Jr, Roberts JE, Hatton DD. Developmental screening and detection of developmental delays in infants and toddlers with fragile X syndrome. J Dev Behav Pediatr. 2004 Feb;25(1):21-7. doi: 10.1097/00004703-200402000-00004. PMID 14767352
- [Background] Carter AS, Volkmar FR, Sparrow SS, Wang JJ, Lord C, Dawson G, Fombonne E, Loveland K, Mesibov G, Schopler E. The Vineland Adaptive Behavior Scales: supplementary norms for individuals with autism. J Autism Dev Disord. 1998 Aug;28(4):287-302. doi: 10.1023/a:1026056518470. PMID 9711485
- [Background] Berry-Kravis E, Krause SE, Block SS, Guter S, Wuu J, Leurgans S, Decle P, Potanos K, Cook E, Salt J, Maino D, Weinberg D, Lara R, Jardini T, Cogswell J, Johnson SA, Hagerman R. Effect of CX516, an AMPA-modulating compound, on cognition and behavior in fragile X syndrome: a controlled trial. J Child Adolesc Psychopharmacol. 2006 Oct;16(5):525-40. doi: 10.1089/cap.2006.16.525. PMID 17069542
- [Background] Wetherby AM, Allen L, Cleary J, Kublin K, Goldstein H. Validity and reliability of the communication and symbolic behavior scales developmental profile with very young children. J Speech Lang Hear Res. 2002 Dec;45(6):1202-18. doi: 10.1044/1092-4388(2002/097). PMID 12546488
- [Background] Picard RW. Future affective technology for autism and emotion communication. Philos Trans R Soc Lond B Biol Sci. 2009 Dec 12;364(1535):3575-84. doi: 10.1098/rstb.2009.0143. PMID 19884152
- [Background] Poh MZ, Swenson NC, Picard RW. A wearable sensor for unobtrusive, long-term assessment of electrodermal activity. IEEE Trans Biomed Eng. 2010 May;57(5):1243-52. doi: 10.1109/TBME.2009.2038487. Epub 2010 Feb 17. PMID 20172811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessments findings during the Screening Visit that could result in ineligibility after informed consent include:
  1. Scoliosis curve > 40º by x-ray
  2. Bone age > 11 years by x-ray
  3. Cardiomegaly by echocardiogram
  4. Tanner Stage II breast development by physical exam
  5. Prolonged QTc by ECG
Groups:
- Placebo First, Then rhIGF-1: One half of subjects will be randomly assigned to receive placebo during the first arm of the study. Subjects assigned to this group will receive twice daily subcutaneous injections of a saline solution (placebo).
- rhIGF-1 First, Then Placebo: One half of subjects will be randomly assigned to receive Recombinant Human Insulin Growth Factor 1 (rhIGF-1) during the first arm of the study. Subjects assigned to this group will receive twice daily subcutaneous injections of IGF-1.
Period: First Intervention (20 Weeks)
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout Period (28 +/- 2 Weeks)
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention (20 Weeks)
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All 30 subjects enrolled and randomized in the study
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rett Syndrome Behavior Questionnaire (RSBQ) - Fear/Anxiety Subscale
Description: The RSBQ is an informant/parent-completed measure of abnormal behaviors typically observed in individuals with RTT, which is completed by a parent/caregiver/LAR. Each item, grouped into eight domains/factors: General mood, Breathing problems, Body rocking and expressionless face, Hand behaviors, Repetitive face movements, Night-time behaviors, Fear/anxiety and Walking/standing), is scored on a Likert scale of 0-2, according to how well the item describes the individual's behavior. A score of "0" indicates the described item is "not true," a score of "1" indicates the described item is "somewhat or sometimes true," and a score of "2" indicates the described item is "very true or often true."
  The total sum of items in each subscale is reported.
  For the fear/anxiety subscale, the sum total could be between 0-8. The higher the sum total score, the greater the frequency of fear/anxiety behaviors.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: In some cases, the number of participants analyzed is less than 15 for each group due to caregiver(s) not completing the forms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 4.00 [3.00 to 6.00] | 5.00 [2.00 to 6.00]
  Visit 2 - First Intervention | 5.00 [3.00 to 6.00] | 3.00 [2.00 to 5.00]
  Visit 3 - First Intervention | 4.00 [3.00 to 5.00] | 3.00 [2.00 to 5.00]
  Visit 4 - First Intervention | 4.00 [2.00 to 5.00] | 3.00 [1.00 to 6.00]
  Visit 5 - First Intervention | 3.00 [2.00 to 5.00] | 3.00 [1.00 to 5.00]
  Visit 6 - Second Intervention | 4.00 [2.00 to 5.00] | 4.00 [2.00 to 6.00]
  Visit 7 - Second Intervention: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention | 4.00 [2.00 to 4.00] | 3.00 [2.00 to 5.00]
  Visit 8 - Second Intervention | 3.00 [3.00 to 5.00] | 4.00 [1.00 to 5.00]
  Visit 9 - Second Intervention | 3.00 [2.00 to 4.00] | 3.00 [1.00 to 5.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention | 4.00 [2.00 to 5.00] | 3.00 [2.00 to 4.00]
  Follow-up: number analyzed (Participants) | 14 | 14
  Follow-up | 3.50 [2.00 to 5.00] | 3.50 [2.00 to 5.00]

2. Primary Outcome: Anxiety, Depression, and Mood Scale (ADAMS) - Social Avoidance Subscale
Description: The ADAMS is completed by the parent/caregiver/LAR and consists of 29 items which are scored on a 4-point rating scale that combines frequency and severity ratings. The instructions ask the rater to describe the individual's behavior over the last six months on the following scale: "0" if the behavior has not occurred, "1" if the behavior occurs occasionally or is a mild problem, "2" if the behavior occurs quite often or is moderate problem, or "3" if the behavior occurs a lot or is a severe problem.
  The Social Avoidance subscale of the ADAMS will be used as a primary outcome measure for this trial. The range for this subscale is 0-21. The higher the subscale score, the more problematic the behavior.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 6.00 [5.00 to 8.00] | 4.00 [2.00 to 8.00]
  Visit 2 - First Intervention | 5.00 [3.00 to 7.00] | 5.00 [3.00 to 7.00]
  Visit 3 - First Intervention | 5.00 [4.00 to 7.00] | 4.00 [2.00 to 7.00]
  Visit 4 - First Intervention | 6.00 [3.00 to 7.00] | 4.00 [3.00 to 7.00]
  Visit 5 - First Intervention | 5.00 [2.00 to 6.00] | 3.00 [2.00 to 5.00]
  Visit 6 - Second Intervention | 4.00 [3.00 to 5.00] | 4.00 [3.00 to 6.00]
  Visit 7 - Second Intervention: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention | 4.00 [2.00 to 7.00] | 4.00 [3.00 to 5.00]
  Visit 8 - Second Intervention | 4.00 [2.00 to 6.00] | 4.00 [3.00 to 5.00]
  Visit 9 - Second Intervention | 3.00 [1.00 to 7.00] | 3.00 [2.00 to 5.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention | 3.50 [2.00 to 5.00] | 3.50 [2.00 to 5.00]
  Follow-up: number analyzed (Participants) | 14 | 14
  Follow-up | 4.00 [2.00 to 6.00] | 3.00 [2.00 to 4.00]

3. Primary Outcome: Clinical Global Impression - Severity (CGI-S)
Description: This scale is used to judge the severity of the subject's disease prior to entry into the study. The clinician will rate the severity of behavioral symptoms at baseline on a 7-point scale from not impaired to the most impaired.
  The scores that correspond to each possible grouping are as follows: 1=Normal, not at all impaired; 2=Borderline impaired; 3=Mildly impaired; 4=Moderately impaired; 5=Markedly impaired; 6=Severely impaired; 7=The most impaired.
  The possible range for reported scores is 1-7.
Time Frame: Every 10 weeks during each of the two 20-week treatment periods
Population: One participant from the "rhIGF-1 First, Then Placebo" group was removed from the study prior to Visit 10, so there is only data for 14 participants included at that time point.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 4.00 [4.00 to 4.00] | 4.00 [3.00 to 4.00]
  Visit 3 - First Intervention | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 4.00]
  Visit 5 - First Intervention | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 5.00]
  Visit 6 - Second Intervention | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 5.00]
  Visit 8 - Second Intervention | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 5.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention | 4.00 [4.00 to 4.00] | 4.50 [4.00 to 5.00]

4. Primary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: Each time the patient was seen after the study intervention was initiated, the clinician compared the patient's overall clinical condition to the CGI-S score obtained at the baseline (visit 1) visit. Based on information collected, the clinician determined if any improvement occurred on the following 7-point scale: 1=Very much improved since the initiation of treatment; 2=Much improved; 3=Minimally improved; 4=No change from baseline (the initiation of treatment); 5=Minimally worse; 6=Much worse; 7=Very much worse since the initiation of treatment.
  The possible range for reported scores is 1-7.
Time Frame: Every 10 weeks during each of the two 20-week treatment periods
Population: Data was not collected at Visit 1 because participants had not yet been exposed to either intervention.
  One participant from the "rhIGF-1 First, Then Placebo" group was removed from the study prior to Visit 10, so there is only data for 14 participants included at that time point.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 3 - First Intervention | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  Visit 5 - First Intervention | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  Visit 6 - Second Intervention | 4.00 [3.00 to 5.00] | 4.00 [4.00 to 5.00]
  Visit 8 - Second Intervention | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 5.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention | 4.00 [3.00 to 4.00] | 4.00 [3.00 to 5.00]

5. Primary Outcome: Parental Global Impression - Severity (PGI-S)
Description: The PGI-S is the parent version of the CGI-S. Parents/caregivers/LAR are asked to rate the severity of their child's symptoms at baseline on a 7-point scale from not at all impaired to the most impaired. The parents/caregivers/LAR will complete the PGI-S at each study visit.
  The scores that correspond to each possible grouping are as follows:
  1=Normal, not at all impaired; 2=Borderline impaired; 3=Mildly impaired; 4=Moderately impaired; 5=Markedly impaired; 6=Severely impaired; 7=The most impaired.
  The possible range for reported scores is 1-7.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 4.00 [3.00 to 4.00] | 6.00 [4.00 to 6.00]
  Visit 2 - First Intervention | 4.00 [3.00 to 6.00] | 4.00 [4.00 to 6.00]
  Visit 3 - First Intervention | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 6.00]
  Visit 4 - First Intervention | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 6.00]
  Visit 5 - First Intervention | 4.00 [4.00 to 6.00] | 4.00 [4.00 to 6.00]
  Visit 6 - Second Intervention | 4.00 [4.00 to 6.00] | 4.00 [4.00 to 6.00]
  Visit 7 - Second Intervention: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 6.00]
  Visit 8 - Second Intervention | 4.00 [4.00 to 4.00] | 6.00 [4.00 to 6.00]
  Visit 9 - Second Intervention | 4.00 [4.00 to 4.00] | 6.00 [4.00 to 6.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention | 4.00 [3.00 to 4.00] | 5.00 [4.00 to 6.00]
  Follow-up: number analyzed (Participants) | 14 | 14
  Follow-up | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 6.00]

6. Primary Outcome: Parental Global Impression - Improvement (PGI-I)
Description: As part of each visit after the study intervention was initiated, the parent/caregiver was asked to compare the patient's overall clinical condition to the score obtained at the baseline (visit 1) visit. Based on information collected, the clinician determined if any improvement occurred on the following 7-point scale: 1=Very much improved since the initiation of treatment; 2=Much improved; 3=Minimally improved; 4=No change from baseline (the initiation of treatment); 5=Minimally worse; 6=Much worse; 7=Very much worse since the initiation of treatment.
  The possible range for reported scores is 1-7.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: Data was not collected at visit 1 because participants had not yet been exposed to either intervention.
  In some cases, the number of participants analyzed is less than 15 for each group due to caregiver(s) not completing the forms.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 2 - First Intervention | 4.00 [3.00 to 4.00] | 4.00 [4.00 to 4.00]
  Visit 3 - First Intervention | 3.00 [3.00 to 4.00] | 4.00 [3.00 to 4.00]
  Visit 4 - First Intervention | 3.00 [3.00 to 4.00] | 4.00 [3.00 to 4.00]
  Visit 5 - First Intervention | 3.00 [3.00 to 4.00] | 3.00 [3.00 to 4.00]
  Visit 6 - Second Intervention | 4.00 [2.00 to 4.00] | 3.00 [3.00 to 4.00]
  Visit 7 - Second Intervention: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention | 3.00 [3.00 to 4.00] | 3.00 [3.00 to 3.00]
  Visit 8 - Second Intervention | 3.00 [3.00 to 4.00] | 3.00 [3.00 to 3.00]
  Visit 9 - Second Intervention | 3.00 [3.00 to 5.00] | 3.00 [3.00 to 3.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention | 3.00 [3.00 to 3.00] | 3.00 [3.00 to 3.00]
  Follow-up: number analyzed (Participants) | 14 | 14
  Follow-up | 3.00 [2.00 to 3.00] | 3.00 [3.00 to 3.00]

7. Primary Outcome: Parent Targeted Visual Analog Scale (PTSVAS) - Scale 1
Description: The parent or caretaker identifies the three most troublesome, RTT-specific, "target" symptoms, such as inattention or breath-holding. This allows the problems that are of concern to parents and the family to be targeted in the trial. In this study the caregiver will choose three target symptoms at baseline and then rate changes in severity of each target symptom on a visual analog scale (VAS).
  The VAS is a 10 cm line, where a target symptom is anchored on one end with the description "the best it has ever been" and on the other with the description "the worst it has ever been." The parent was asked to marked on the line where they felt their child's symptoms currently fit best. This mark was measured as recorded as a numeric value from 0.00-10.00 cm. The higher the value, the worse the symptom.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 6.50 [3.25 to 8.40] | 8.80 [5.05 to 9.85]
  Visit 2 - First Intervention: number analyzed (Participants) | 13 | 13
  Visit 2 - First Intervention | 4.70 [3.45 to 7.70] | 4.80 [2.30 to 8.95]
  Visit 3 - First Intervention | 5.65 [3.55 to 8.90] | 5.35 [3.80 to 9.35]
  Visit 4 - First Intervention: number analyzed (Participants) | 11 | 11
  Visit 4 - First Intervention | 5.05 [2.55 to 7.70] | 5.10 [4.80 to 9.10]
  Visit 5 - First Intervention | 4.80 [2.00 to 7.50] | 5.15 [2.90 to 9.55]
  Visit 6 - Second Intervention: number analyzed (Participants) | 14 | 15
  Visit 6 - Second Intervention | 4.95 [3.75 to 8.50] | 5.20 [4.70 to 9.25]
  Visit 7 - Second Intervention: number analyzed (Participants) | 11 | 13
  Visit 7 - Second Intervention | 4.55 [2.55 to 6.00] | 4.65 [3.85 to 7.25]
  Visit 8 - Second Intervention | 5.65 [3.70 to 7.55] | 5.00 [3.65 to 7.45]
  Visit 9 - Second Intervention: number analyzed (Participants) | 13 | 12
  Visit 9 - Second Intervention | 4.15 [2.45 to 6.45] | 5.15 [3.63 to 8.58]
  Visit 10 - Second Intervention: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention | 4.80 [2.50 to 6.90] | 5.05 [4.20 to 8.50]
  Follow-up: number analyzed (Participants) | 9 | 12
  Follow-up | 5.60 [1.40 to 6.25] | 5.08 [4.13 to 8.13]

8. Primary Outcome: Parent Targeted Visual Analog Scale (PTSVAS) - Scale 2
Description: as for outcome 7
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 7.75 [4.80 to 9.45] | 6.35 [5.20 to 9.85]
  Visit 2 - First Intervention | 4.50 [3.75 to 5.00] | 5.25 [4.85 to 8.40]
  Visit 3 - First Intervention | 5.85 [4.30 to 7.25] | 5.95 [4.95 to 8.90]
  Visit 4 - First Intervention | 5.00 [3.05 to 6.20] | 5.40 [4.90 to 6.45]
  Visit 5 - First Intervention | 5.00 [3.30 to 6.10] | 5.45 [1.40 to 7.80]
  Visit 6 - Second Intervention | 5.35 [4.95 to 7.85] | 7.10 [4.95 to 9.25]
  Visit 7 - Second Intervention | 5.50 [3.85 to 6.20] | 5.85 [3.40 to 6.90]
  Visit 8 - Second Intervention | 5.15 [3.80 to 7.20] | 5.00 [3.00 to 7.60]
  Visit 9 - Second Intervention | 3.80 [1.70 to 6.35] | 5.13 [3.43 to 7.05]
  Visit 10 - Second Intervention | 4.90 [2.60 to 6.80] | 4.95 [2.25 to 8.15]
  Follow-up | 5.15 [3.85 to 6.65] | 5.20 [3.60 to 7.95]

9. Primary Outcome: Parent Targeted Visual Analog Scale (PTSVAS) - Scale 3
Description: as for outcome 7
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 7.85 [5.70 to 8.70] | 5.70 [4.50 to 9.65]
  Visit 2 - First Intervention: number analyzed (Participants) | 12 | 13
  Visit 2 - First Intervention | 4.70 [4.48 to 8.30] | 5.00 [2.55 to 5.40]
  Visit 3 - First Intervention | 5.65 [3.65 to 9.00] | 5.20 [3.50 to 9.40]
  Visit 4 - First Intervention: number analyzed (Participants) | 11 | 11
  Visit 4 - First Intervention | 4.15 [2.90 to 6.05] | 5.35 [3.50 to 8.65]
  Visit 5 - First Intervention | 5.00 [4.40 to 7.40] | 5.10 [4.00 to 8.20]
  Visit 6 - Second Intervention: number analyzed (Participants) | 14 | 15
  Visit 6 - Second Intervention | 6.20 [4.70 to 8.35] | 5.35 [4.05 to 9.05]
  Visit 7 - Second Intervention: number analyzed (Participants) | 11 | 13
  Visit 7 - Second Intervention | 4.80 [3.15 to 7.30] | 4.95 [2.95 to 7.05]
  Visit 8 - Second Intervention | 4.85 [3.80 to 8.15] | 5.15 [1.75 to 7.10]
  Visit 9 - Second Intervention: number analyzed (Participants) | 13 | 12
  Visit 9 - Second Intervention | 4.60 [3.15 to 7.90] | 5.25 [3.35 to 7.10]
  Visit 10 - Second Intervention: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention | 4.13 [1.10 to 8.45] | 4.55 [2.95 to 5.45]
  Follow-up: number analyzed (Participants) | 9 | 12
  Follow-up | 4.55 [2.20 to 7.00] | 5.10 [3.20 to 8.03]

10. Primary Outcome: Kerr Clinical Severity Scale
Description: The Kerr clinical severity scale (Kerr scale) is a quantitative measure of global disease severity. The Kerr scale is a summation of individual items related to Rett syndrome phenotypic characteristics. The items are based on the severity or degree of abnormality of each characteristic on a discrete scale (0, 1, 2) with the highest level corresponding to the most severe or most abnormal presentations.
  The possible range of scores is 0-48. The higher the score, the more severe the symptoms.
Time Frame: At the start and end of each 20-week treatment period
Population: In some cases, the number of participants analyzed is less than 15 for each group due to caregiver(s) not completing the forms.
  One participant from the "rhIGF-1 First, Then Placebo" group was removed from the study prior to Visit 10, so there is only data for 14 participants included at that time point.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention | 16.50 [13.00 to 20.00] | 18.00 [12.00 to 22.00]
  Visit 5 - First Intervention | 15.00 [13.00 to 21.00] | 18.00 [14.00 to 22.00]
  Visit 6 - Second Intervention | 15.00 [12.00 to 20.00] | 19.00 [16.00 to 22.00]
  Visit 10 - Second Intervention: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention | 14.00 [13.00 to 22.00] | 20.00 [17.00 to 22.00]

11. Secondary Outcome: Rett Syndrome Behavior Questionnaire (RSBQ)
Description: The RSBQ is a parent-completed measure of abnormal behaviors typically observed in individuals with RTT. Each item, grouped into eight subscales, is scored on a Likert scale of 0-2, according to how well the item describes the individual's behavior. A score of "0" indicates the described item is "not true," a score of "1" indicates the described item is "somewhat or sometimes true," and a score of "2" indicates the described item is "very true or often true."
  The total sum of each subscale is reported. The higher the score, the more severe the symptoms of that subscale in the participant.
  The range for each subscale is as follows:
  General Mood: 0-16 Body rocking and expressionless face: 0-14 Hand behaviors: 0-12 Breathing Problems: 0-10 Repetitive Face Movements: 0-8 Night-time behaviors: 0-6 Walking Standing: 0-4
  The fear/anxiety subscale was used as a primary outcome measure in this study and results can be found in that section.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1- First Intervention: General Mood | 7.00 [4.00 to 11.00] | 4.00 [3.00 to 7.00]
  Visit 2- First Intervention: General Mood | 5.00 [3.00 to 8.00] | 3.00 [1.00 to 4.00]
  Visit 3- First Intervention: General Mood | 6.00 [1.00 to 8.00] | 2.00 [1.00 to 4.00]
  Visit 4- First Intervention: General Mood | 5.00 [3.00 to 8.00] | 2.00 [1.00 to 5.00]
  Visit 5- First Intervention: General Mood | 5.00 [1.00 to 8.00] | 3.00 [1.00 to 6.00]
  Visit 6- Second Intervention: General Mood | 4.00 [2.00 to 8.00] | 4.00 [2.00 to 6.00]
  Visit 7- Second Intervention: General Mood: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: General Mood | 5.50 [2.00 to 7.00] | 2.00 [1.00 to 5.00]
  Visit 8- Second Intervention: General Mood | 5.00 [2.00 to 8.00] | 2.00 [1.00 to 4.00]
  Visit 9- Second Intervention: General Mood | 6.00 [3.00 to 8.00] | 1.00 [1.00 to 5.00]
  Visit 10- Second Intervention: General Mood: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: General Mood | 4.00 [2.00 to 8.00] | 2.50 [1.00 to 6.00]
  Follow-up: General Mood: number analyzed (Participants) | 14 | 14
  Follow-up: General Mood | 5.50 [3.00 to 6.00] | 2.00 [1.00 to 4.00]
  Visit 1- First Intervention: Body Rocking | 6.00 [5.00 to 10.00] | 4.00 [4.00 to 6.00]
  Visit 2- First Intervention: Body Rocking | 5.00 [4.00 to 7.00] | 4.00 [3.00 to 6.00]
  Visit 3- First Intervention: Body Rocking | 5.00 [3.00 to 8.00] | 3.00 [2.00 to 6.00]
  Visit 4- First Intervention: Body Rocking | 6.00 [4.00 to 7.00] | 4.00 [2.00 to 5.00]
  Visit 5- First Intervention: Body Rocking | 5.00 [3.00 to 8.00] | 4.00 [2.00 to 5.00]
  Visit 6- Second Intervention: Body Rocking | 4.00 [3.00 to 7.00] | 4.00 [3.00 to 5.00]
  Visit 7- Second Intervention: Body Rocking: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Body Rocking | 5.00 [3.00 to 7.00] | 3.00 [3.00 to 5.00]
  Visit 8- Second Intervention: Body Rocking | 5.00 [3.00 to 6.00] | 4.00 [2.00 to 5.00]
  Visit 9- Second Intervention: Body Rocking | 4.00 [3.00 to 7.00] | 3.00 [2.00 to 5.00]
  Visit 10- Second Intervention: Body Rocking: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Body Rocking | 5.00 [3.00 to 7.00] | 4.00 [2.00 to 5.00]
  Followup: Body Rocking: number analyzed (Participants) | 14 | 14
  Followup: Body Rocking | 4.50 [3.00 to 7.00] | 4.00 [2.00 to 5.00]
  Visit 1- First Intervention: Hand Behaviors | 8.00 [7.00 to 10.00] | 8.00 [5.00 to 10.00]
  Visit 2- First Intervention: Hand Behaviors | 9.00 [6.00 to 9.00] | 8.00 [6.00 to 10.00]
  Visit 3- First Intervention: Hand Behaviors | 8.00 [7.00 to 10.00] | 8.00 [5.00 to 9.00]
  Visit 4- First Intervention: Hand Behaviors | 8.00 [6.00 to 9.00] | 9.00 [6.00 to 9.00]
  Visit 5- First Intervention: Hand Behaviors | 8.00 [6.00 to 10.00] | 9.00 [5.00 to 10.00]
  Visit 6- Second Intervention: Hand Behaviors | 9.00 [6.00 to 10.00] | 8.00 [7.00 to 10.00]
  Visit 7- Second Intervention: Hand Behaviors: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Hand Behaviors | 8.00 [5.00 to 10.00] | 9.00 [6.00 to 9.00]
  Visit 8- Second Intervention: Hand Behaviors | 8.00 [6.00 to 9.00] | 9.00 [6.00 to 9.00]
  Visit 9- Second Intervention: Hand Behaviors | 8.00 [5.00 to 9.00] | 7.00 [6.00 to 10.00]
  Visit 10- Second Intervention: Hand Behaviors: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Hand Behaviors | 7.00 [6.00 to 9.00] | 9.00 [6.00 to 10.00]
  Follow-up: Hand Behaviors: number analyzed (Participants) | 14 | 14
  Follow-up: Hand Behaviors | 7.50 [7.00 to 9.00] | 8.50 [6.00 to 10.00]
  Visit 1- First Intervention: Breathing Problems | 6.00 [3.00 to 9.00] | 4.00 [3.00 to 7.00]
  Visit 2- First Intervention: Breathing Problems | 4.00 [2.00 to 8.00] | 4.00 [2.00 to 6.00]
  Visit 3- First Intervention: Breathing Problems | 5.00 [2.00 to 8.00] | 4.00 [2.00 to 6.00]
  Visit 4- First Intervention: Breathing Problems | 5.00 [3.00 to 7.00] | 5.00 [2.00 to 7.00]
  Visit 5- First Intervention: Breathing Problems | 5.00 [1.00 to 8.00] | 4.00 [2.00 to 7.00]
  Visit 6- Second Intervention: Breathing Problems | 6.00 [2.00 to 9.00] | 4.00 [1.00 to 8.00]
  Visit 7- Second Intervention: Breathing Problems: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Breathing Problems | 4.50 [2.00 to 7.00] | 3.00 [1.00 to 7.00]
  Visit 8- Second Intervention: Breathing Problems | 6.00 [3.00 to 7.00] | 3.00 [1.00 to 6.00]
  Visit 9- Second Intervention: Breathing Problems | 5.00 [2.00 to 7.00] | 3.00 [0.00 to 5.00]
  Visit 10- Second Intervention: Breathing Problems: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Breathing Problems | 6.00 [3.00 to 7.00] | 4.00 [1.00 to 5.00]
  Follow-up: Breathing Problems: number analyzed (Participants) | 14 | 14
  Follow-up: Breathing Problems | 5.00 [2.00 to 7.00] | 3.00 [0.00 to 4.00]
  Visit 1- First Intervention: Repetitive Face Movem | 2.00 [1.00 to 5.00] | 2.00 [2.00 to 4.00]
  Visit 2- First Intervention: Repetitive Face Movem | 2.00 [0.00 to 4.00] | 2.00 [2.00 to 4.00]
  Visit 3- First Intervention: Repetitive Face Movem | 3.00 [1.00 to 4.00] | 3.00 [2.00 to 4.00]
  Visit 4- First Intervention: Repetitive Face Movem | 2.00 [1.00 to 5.00] | 2.00 [1.00 to 4.00]
  Visit 5- First Intervention: Repetitive Face Movem | 3.00 [0.00 to 5.00] | 2.00 [0.00 to 4.00]
  Visit 6- Second Intervention: Repetitive Face Mov | 3.00 [2.00 to 5.00] | 3.00 [2.00 to 4.00]
  Visit 7- Second Intervention: Repetitive Face Mov: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Repetitive Face Mov | 3.00 [1.00 to 5.00] | 2.00 [0.00 to 4.00]
  Visit 8- Second Intervention: Repetitive Face Mov | 3.00 [2.00 to 4.00] | 2.00 [1.00 to 4.00]
  Visit 9- Second Intervention: Repetitive Face Mov | 3.00 [1.00 to 5.00] | 2.00 [0.00 to 3.00]
  Visit 10- Second Intervention: Repetitive Face Mov: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Repetitive Face Mov | 3.00 [1.00 to 5.00] | 1.50 [1.00 to 4.00]
  Follow-up: Repetitive Face Movements: number analyzed (Participants) | 14 | 14
  Follow-up: Repetitive Face Movements | 2.00 [1.00 to 4.00] | 2.00 [0.00 to 2.00]
  Visit 1- First Intervention: Night time Behaviors | 0.00 [0.00 to 2.00] | 1.00 [0.00 to 2.00]
  Visit 2- First Intervention: Night time Behaviors | 0.00 [0.00 to 3.00] | 1.00 [0.00 to 2.00]
  Visit 3- First Intervention: Night time Behaviors | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 2.00]
  Visit 4- First Intervention: Night time Behaviors | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00]
  Visit 5- First Intervention: Night time Behaviors | 0.00 [0.00 to 2.00] | 1.00 [0.00 to 2.00]
  Visit 6- Second Intervention: Night time Behavior | 0.00 [0.00 to 2.00] | 1.00 [0.00 to 2.00]
  Visit 7- Second Intervention: Night time Behavior: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Night time Behavior | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00]
  Visit 8- Second Intervention: Night time Behavior | 1.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00]
  Visit 9- Second Intervention: Night time Behavior | 0.00 [0.00 to 3.00] | 0.00 [0.00 to 1.00]
  Visit 10- Second Intervention: Night time Behavior: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Night time Behavior | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00]
  Follow-up: Night time Behaviors: number analyzed (Participants) | 14 | 14
  Follow-up: Night time Behaviors | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00]
  Visit 1- First Intervention: Walking/Standing | 2.00 [2.00 to 3.00] | 2.00 [1.00 to 3.00]
  Visit 2- First Intervention: Walking/Standing | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00]
  Visit 3- First Intervention: Walking/Standing | 2.00 [2.00 to 2.00] | 2.00 [1.00 to 3.00]
  Visit 4- First Intervention: Walking/Standing | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00]
  Visit 5- First Intervention: Walking/Standing | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00]
  Visit 6- Second Intervention: Walking/Standing | 2.00 [2.00 to 3.00] | 2.00 [1.00 to 2.00]
  Visit 7- Second Intervention: Walking/Standing: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Walking/Standing | 2.00 [2.00 to 3.00] | 2.00 [1.00 to 3.00]
  Visit 8- Second Intervention: Walking/Standing | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00]
  Visit 9- Second Intervention: Walking/Standing | 3.00 [1.00 to 3.00] | 2.00 [1.00 to 2.00]
  Visit 10- Second Intervention: Walking/Standing: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Walking/Standing | 1.50 [1.00 to 3.00] | 2.00 [1.00 to 2.00]
  Follow-up: Walking/Standing: number analyzed (Participants) | 14 | 14
  Follow-up: Walking/Standing | 2.00 [1.00 to 3.00] | 2.00 [2.00 to 3.00]

12. Secondary Outcome: Anxiety, Depression, and Mood Scale (ADAMS)
Description: Remaining subscales of the ADAMS that are not primary outcome measures include: Manic/hyperactive, Depressed mood, General anxiety, Obsessive/compulsive behavior.
  The range for each subscale is as follows:
  Manic/Hyperactive Behavior: 0-15 Depressed Mood: 0-21 General Anxiety: 0-21 Obsessive/Compulsive Behavior: 0-9
  The higher the score for each subscale, the more problematic the behavior.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1- First Intervention: Manic/Hyperactive | 8.00 [5.00 to 11.00] | 7.00 [5.00 to 9.00]
  Visit 2- First Intervention: Manic/Hyperactive | 7.00 [3.00 to 10.00] | 7.00 [4.00 to 9.00]
  Visit 3- First Intervention: Manic/Hyperactive | 7.00 [3.00 to 9.00] | 6.00 [4.00 to 7.00]
  Visit 4- First Intervention: Manic/Hyperactive | 7.00 [5.00 to 9.00] | 5.00 [4.00 to 7.00]
  Visit 5- First Intervention: Manic/Hyperactive | 7.00 [4.00 to 9.00] | 4.00 [3.00 to 7.00]
  Visit 6- Second Intervention: Manic/Hyperactive | 8.00 [3.00 to 9.00] | 6.00 [5.00 to 8.00]
  Visit 7- Second Intervention: Manic/Hyperactive: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Manic/Hyperactive | 6.50 [3.00 to 9.00] | 5.00 [3.00 to 7.00]
  Visit 8- Second Intervention: Manic/Hyperactive | 6.00 [3.00 to 8.00] | 5.00 [3.00 to 6.00]
  Visit 9- Second Intervention: Manic/Hyperactive | 6.00 [4.00 to 9.00] | 4.00 [1.00 to 6.00]
  Visit 10- First Intervention: Manic/Hyperactive: number analyzed (Participants) | 14 | 14
  Visit 10- First Intervention: Manic/Hyperactive | 5.00 [2.00 to 7.00] | 4.50 [2.00 to 7.00]
  Follow-up: Manic/Hyperactive Subscale: number analyzed (Participants) | 14 | 14
  Follow-up: Manic/Hyperactive Subscale | 5.00 [3.00 to 9.00] | 5.00 [3.00 to 7.00]
  Visit 1- First Intervention: Depressed Mood | 2.00 [2.00 to 7.00] | 4.00 [3.00 to 6.00]
  Visit 2- First Intervention: Depressed Mood | 4.00 [1.00 to 5.00] | 5.00 [2.00 to 6.00]
  Visit 3- First Intervention: Depressed Mood | 3.00 [1.00 to 5.00] | 3.00 [2.00 to 5.00]
  Visit 4- First Intervention: Depressed Mood | 2.00 [1.00 to 4.00] | 3.00 [1.00 to 5.00]
  Visit 5- First Intervention: Depressed Mood | 2.00 [1.00 to 4.00] | 4.00 [0.00 to 5.00]
  Visit 6- Second Intervention: Depressed Mood | 2.00 [0.00 to 5.00] | 4.00 [3.00 to 6.00]
  Visit 7- Second Intervention: Depressed Mood: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Depressed Mood | 3.00 [0.00 to 6.00] | 3.00 [2.00 to 5.00]
  Visit 8- Second Intervention: Depressed Mood | 2.00 [1.00 to 5.00] | 3.00 [1.00 to 5.00]
  Visit 9- Second Intervention: Depressed Mood | 3.00 [0.00 to 4.00] | 2.00 [1.00 to 5.00]
  Visit 10- Second Intervention: Depressed Mood: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: Depressed Mood | 2.00 [1.00 to 4.00] | 3.00 [2.00 to 4.00]
  Follow-up: Depressed Mood Subscale: number analyzed (Participants) | 14 | 14
  Follow-up: Depressed Mood Subscale | 2.00 [0.00 to 5.00] | 3.50 [0.00 to 4.00]
  Visit 1- First Intervention: General Anxiety | 8.00 [5.00 to 12.00] | 6.00 [5.00 to 12.00]
  Visit 2- First Intervention: General Anxiety | 6.00 [4.00 to 12.00] | 7.00 [3.00 to 10.00]
  Visit 3- First Intervention: General Anxiety | 6.00 [3.00 to 9.00] | 6.00 [3.00 to 9.00]
  Visit 4- First Intervention: General Anxiety | 5.00 [2.00 to 11.00] | 5.00 [2.00 to 8.00]
  Visit 5- First Intervention: General Anxiety | 5.00 [2.00 to 10.00] | 5.00 [3.00 to 7.00]
  Visit 6- Second Intervention: General Anxiety | 6.00 [3.00 to 9.00] | 7.00 [3.00 to 11.00]
  Visit 7- Second Intervention: General Anxiety: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: General Anxiety | 6.00 [2.00 to 8.00] | 5.00 [1.00 to 7.00]
  Visit 8- Second Intervention: General Anxiety | 6.00 [3.00 to 9.00] | 4.00 [2.00 to 8.00]
  Visit 9- Second Intervention: General Anxiety | 4.00 [2.00 to 8.00] | 3.00 [1.00 to 6.00]
  Visit 10- Second Intervention: General Anxiety: number analyzed (Participants) | 14 | 14
  Visit 10- Second Intervention: General Anxiety | 4.00 [2.00 to 7.00] | 4.00 [2.00 to 5.00]
  Follow-up: General Anxiety Subscale: number analyzed (Participants) | 14 | 14
  Follow-up: General Anxiety Subscale | 5.50 [3.00 to 9.00] | 4.00 [1.00 to 6.00]
  Visit 1- First Intervention: Obsessive Compulsive | 4.00 [3.00 to 6.00] | 3.00 [0.00 to 5.00]
  Visit 2- First Intervention: Obsessive Compulsive | 4.00 [2.00 to 4.00] | 4.00 [1.00 to 4.00]
  Visit 3- First Intervention: Obsessive Compulsive | 4.00 [1.00 to 4.00] | 4.00 [1.00 to 4.00]
  Visit 4- First Intervention: Obsessive Compulsive | 3.00 [3.00 to 4.00] | 3.00 [1.00 to 4.00]
  Visit 5- First Intervention: Obsessive Compulsive | 3.00 [2.00 to 4.00] | 3.00 [0.00 to 4.00]
  Visit 6- Second Intervention: Obsessive Compulsive | 3.00 [1.00 to 5.00] | 3.00 [1.00 to 5.00]
  Visit 7- Second Intervention: Obsessive Compulsive: number analyzed (Participants) | 14 | 15
  Visit 7- Second Intervention: Obsessive Compulsive | 3.00 [2.00 to 6.00] | 3.00 [0.00 to 4.00]
  Visit 8- Second Intervention: Obsessive Compulsive | 3.00 [2.00 to 4.00] | 3.00 [0.00 to 4.00]
  Visit 9- Second Intervention: Obsessive Compulsive | 3.00 [1.00 to 3.00] | 2.00 [0.00 to 4.00]
  Visit 10- First Intervention: Obsessive Compulsive: number analyzed (Participants) | 14 | 14
  Visit 10- First Intervention: Obsessive Compulsive | 2.00 [1.00 to 4.00] | 2.50 [0.00 to 5.00]
  Follow-up: Obsessive Compulsive Behavior Subscale: number analyzed (Participants) | 14 | 14
  Follow-up: Obsessive Compulsive Behavior Subscale | 3.50 [2.00 to 4.00] | 3.00 [0.00 to 4.00]

13. Secondary Outcome: Mullen Scales of Early Learning (MSEL)
Description: The MSEL is a standardized developmental test for children ages 3 to 68 months consisting of five subscales: gross motor, fine motor, visual reception, expressive language, and receptive language.
  The raw score is reported for each subscale domain. The potential score ranges are as follows:
  Visual Reception: 33 items, score range=0-50, Fine Motor: 30 items, score range= 0-49, Receptive Language: 33 items, score range= 0-48, Expressive Language: 28 items, score range= 0-50. The gross motor subscale was not included in this population.
  A higher raw score indicates more advanced abilities in that section.
Time Frame: At the start and end of each 20-week treatment period
Population: One participant from the "rhIGF-1 First, Then Placebo" group was removed from the study prior to Visit 10, so there is only data for 14 participants included at that time point.
  In some cases, the number of participants analyzed is less than 15 for each group due to subject's inability or unwillingness to complete the testing.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1- First Intervention: Visual Reception | 17.00 [15.00 to 25.00] | 26.00 [18.00 to 42.00]
  Visit 5- First Intervention: Visual Reception: number analyzed (Participants) | 15 | 14
  Visit 5- First Intervention: Visual Reception | 26.00 [16.00 to 33.00] | 39.50 [20.00 to 49.00]
  Visit 6- Second Intervention: Visual Reception | 23.00 [20.00 to 36.00] | 42.00 [23.00 to 48.00]
  Visit 10: Visual Reception Raw Score: number analyzed (Participants) | 15 | 13
  Visit 10: Visual Reception Raw Score | 28.00 [25.00 to 41.00] | 44.00 [28.00 to 48.00]
  Visit 1- First Intervention: Fine Motor | 10.00 [7.00 to 14.00] | 7.00 [6.00 to 17.00]
  Visit 5- First Intervention: Fine Motor | 9.00 [6.00 to 13.00] | 7.00 [3.00 to 15.00]
  Visit 6- Second Intervention: Fine Motor | 11.00 [7.00 to 13.00] | 10.00 [5.00 to 17.00]
  Visit 10- Second Intervention: Fine Motor: number analyzed (Participants) | 15 | 14
  Visit 10- Second Intervention: Fine Motor | 9.00 [6.00 to 13.00] | 8.50 [4.00 to 13.00]
  Visit 1- First Intervention: Receptive Language: number analyzed (Participants) | 15 | 14
  Visit 1- First Intervention: Receptive Language | 20.00 [17.00 to 31.00] | 25.50 [17.00 to 40.00]
  Visit 5- First Intervention: Receptive Language | 30.00 [19.00 to 33.00] | 32.00 [25.00 to 44.00]
  Visit 6- Second Intervention: Receptive Language | 31.00 [24.00 to 35.00] | 38.00 [33.00 to 47.00]
  Visit 10- Second Intervention: Receptive Language: number analyzed (Participants) | 15 | 14
  Visit 10- Second Intervention: Receptive Language | 31.00 [26.00 to 38.00] | 36.50 [27.00 to 44.00]
  Visit 1- First Intervention: Expressive Language | 8.00 [5.00 to 9.00] | 9.00 [6.00 to 11.00]
  Visit 5- First Intervention: Expressive Language | 9.00 [5.00 to 11.00] | 8.00 [5.00 to 11.00]
  Visit 6- Second Intervention: Expressive Language | 6.00 [5.00 to 9.00] | 10.00 [5.00 to 12.00]
  Visit 10- Second Intervention: Expressive Language: number analyzed (Participants) | 15 | 14
  Visit 10- Second Intervention: Expressive Language | 8.00 [5.00 to 10.00] | 8.00 [6.00 to 12.00]

14. Secondary Outcome: Vineland Adaptive Behavior Scales, Second Edition (VABS-II)
Description: The VABS-II is a survey designed to assess personal and social functioning. Within each domain (Communication, Daily Living Skills, Socialization, and Motor Skills), items can given a score of "2" if the participant successfully performs the activity usually; a "1" if the participant successfully performs the activity sometimes, or needs reminders; a "0" if the participant never performs the activity, and a "DK" if the parent/caregiver is unsure of the participant's ability for an item.
  The raw scores in each sub-domain are reported and the ranges for these are as follows: [Communication Domain], Receptive Language=0-40, Expressive Language=0-108, Written Language=0-50; [Daily Living Skills Domain], Personal=0-82, Domestic=0-48, Community=0-88; [Socialization Domain], Interpersonal Relationships=0-76, Play and Leisure Time=0-62, Coping Skills=0-60; [Motor Skills Domain]: Gross Motor Skills=0-80, Fine Motor Skills=0-72.
  A higher score indicates more advanced abilities.
Time Frame: At the start and end of each 20-week treatment period
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention: Receptive | 13.00 [9.00 to 16.00] | 18.00 [13.00 to 20.00]
  Visit 5 - First Intervention: Receptive | 15.00 [14.00 to 20.00] | 21.00 [17.00 to 23.00]
  Visit 6 - Second Intervention: Receptive Language: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Receptive Language | 18.00 [13.00 to 20.00] | 22.00 [20.00 to 24.00]
  Visit 10 - Second Intervention: Receptive Language: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Receptive Language | 20.00 [15.00 to 24.00] | 24.50 [20.00 to 29.00]
  Visit 1 - First Intervention: Expressive | 16.00 [12.00 to 17.00] | 18.00 [13.00 to 25.00]
  Visit 5 - First Intervention: Expressive | 17.00 [13.00 to 23.00] | 22.00 [18.00 to 29.00]
  Visit 6 - Second Intervention: Expressive Lang.: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Expressive Lang. | 18.00 [11.00 to 23.00] | 25.00 [18.00 to 31.00]
  Visit 10 - Second Intervention: Expressive Lang.: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Expressive Lang. | 20.00 [15.00 to 28.00] | 24.00 [23.00 to 34.0]
  Visit 1 - First Intervention: Written | 0.00 [0.00 to 1.00] | 4.00 [0.00 to 7.00]
  Visit 5 - First Intervention: Written | 0.00 [0.00 to 5.00] | 5.00 [0.00 to 9.00]
  Visit 6: - Second Intervention Written Language: number analyzed (Participants) | 15 | 14
  Visit 6: - Second Intervention Written Language | 4.00 [1.00 to 7.00] | 7.00 [2.00 to 9.00]
  Visit 10 - Second Intervention: Written Language: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Written Language | 6.00 [0.00 to 8.00] | 7.00 [4.00 to 10.00]
  Visit 1 - First Intervention: Personal | 9.00 [7.00 to 10.00] | 8.00 [6.00 to 10.00]
  Visit 5 - First Intervention: Personal | 10.00 [8.00 to 13.00] | 9.00 [7.00 to 13.00]
  Visit 6 - Second Intervention: Personal: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Personal | 9.00 [8.00 to 14.00] | 8.50 [8.00 to 16.00]
  Visit 10 - Second Intervention: Personal: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Personal | 10.00 [7.00 to 14.00] | 9.50 [8.00 to 10.00]
  Visit 1 - First Intervention: Domestic | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00]
  Visit 5 - First Intervention: Domestic | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00]
  Visit 6 - Second Intervention: Domestic: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Domestic | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 2.00]
  Visit 10 - Second Intervention: Domestic: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Domestic | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00]
  Visit 1 - First Intervention: Community | 0.00 [0.00 to 1.00] | 3.00 [2.00 to 6.00]
  Visit 5 - First Intervention: Community | 1.00 [0.00 to 2.00] | 3.00 [2.00 to 4.00]
  Visit 6 - Second Intervention: Community: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Community | 1.00 [0.00 to 3.00] | 5.00 [2.00 to 7.00]
  Visit 10 - Second Intervention: Community: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Community | 2.00 [0.00 to 5.00] | 5.00 [2.00 to 7.00]
  Visit 1 - First Intervention: Interpersonal Rel. | 18.00 [15.00 to 21.00] | 21.00 [17.00 to 24.00]
  Visit 5 - First Intervention: Interpersonal Rel. | 18.00 [15.00 to 21.00] | 22.00 [17.00 to 25.00]
  Visit 6 - Second Intervention: Interpersonal Rel.: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Interpersonal Rel. | 19.00 [15.00 to 21.00] | 21.00 [20.00 to 26.00]
  Visit 10 - Second Intervention: Interpersonal Rel.: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Interpersonal Rel. | 20.00 [16.00 to 23.00] | 22.50 [19.00 to 27.00]
  Visit 1 - First Intervention: Play and Leisure | 8.00 [7.00 to 12.00] | 13.00 [11.00 to 17.00]
  Visit 5 - First Intervention: Play and Leisure | 11.00 [9.00 to 12.00] | 12.00 [11.00 to 16.00]
  Visit 6 - Second Intervention: Play and Leisure: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Play and Leisure | 12.00 [9.00 to 14.00] | 13.00 [11.00 to 16.00]
  Visit 10 - Second Intervention: Play and Leisure: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Play and Leisure | 11.00 [9.00 to 15.00] | 12.50 [10.00 to 16.00]
  Visit 1 - First Intervention: Coping Skills | 3.00 [2.00 to 4.00] | 3.00 [3.00 to 4.00]
  Visit 5 - First Intervention: Coping Skills | 2.00 [2.00 to 4.00] | 4.00 [2.00 to 6.00]
  Visit 6 - Second Intervention: Coping Skills: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Coping Skills | 3.00 [3.00 to 4.00] | 6.00 [3.00 to 6.00]
  Visit 10 - Second Intervention: Coping Skills: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Coping Skills | 4.00 [3.00 to 5.00] | 4.50 [3.00 to 8.00]
  Visit 1 - First Intervention: Gross Motor | 31.00 [21.00 to 37.00] | 10.00 [7.00 to 43.00]
  Visit 5 - First Intervention: Gross Motor | 34.00 [22.00 to 42.00] | 10.00 [8.00 to 36.00]
  Visit 6 - Second Intervention: Gross Motor: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Gross Motor | 27.00 [12.00 to 45.00] | 11.50 [8.00 to 34.00]
  Visit 10 - Second Intervention: Gross Motor: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Gross Motor | 27.00 [14.00 to 46.00] | 10.50 [8.00 to 30.00]
  Visit 1 - First Intervention: Fine Motor | 6.00 [3.00 to 8.00] | 2.00 [1.00 to 14.00]
  Visit 5 - First Intervention: Fine Motor | 6.00 [4.00 to 9.00] | 3.00 [2.00 to 15.00]
  Visit 6 - Second Intervention: Fine Motor: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Fine Motor | 7.00 [3.00 to 10.00] | 4.00 [2.00 to 16.00]
  Visit 10 - Second Intervention: Fine Motor: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Fine Motor | 5.00 [2.00 to 9.00] | 4.00 [2.00 to 8.00]

15. Secondary Outcome: Communication and Symbolic Behavior Scales - Developmental Profile (CSBS-DP)
Description: The CSBS-DP was designed to measure early communication and symbolic skills in infants and young children (that is, functional communication skills of 6 month to 2 year olds). The CSBS-DP measures skills from three composites: (a) Social (emotion, eye gaze, and communication); (b) Speech (sounds and words); and (c) Symbolic (understanding and object use) and asks about developmental milestones. The data reported are the composite scores for these three categories.
  The possible scores for the three composite categories are as follows:
  Social Composite = 0-48; Speech Composite = 0-40; Symbolic Composite = 0-51.
  A higher score indicates more advanced abilities in that area.
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention: Social | 19.00 [16.00 to 25.00] | 22.00 [19.00 to 26.00]
  Visit 2: Social Composite Score | 20.00 [15.00 to 23.00] | 24.00 [20.00 to 28.00]
  Visit 3: Social Composite Score | 18.00 [13.00 to 25.00] | 24.00 [21.00 to 30.00]
  Visit 4: Social Composite Score | 18.00 [17.00 to 25.00] | 24.00 [21.00 to 31.00]
  Visit 5: Social Composite Score | 20.00 [15.00 to 29.00] | 23.00 [21.00 to 34.00]
  Visit 6 - Second Intervention: Social | 18.00 [15.00 to 28.00] | 28.00 [22.00 to 34.00]
  Visit 7 - Second Intervention: Social: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention: Social | 20.00 [16.00 to 26.00] | 25.00 [21.00 to 34.00]
  Visit 8 - Second Intervention: Social: number analyzed (Participants) | 15 | 14
  Visit 8 - Second Intervention: Social | 21.00 [17.00 to 27.00] | 27.00 [25.00 to 36.00]
  Visit 9 - Second Intervention: Social | 21.00 [17.00 to 29.00] | 29.00 [25.00 to 34.00]
  Visit 10 - Second Intervention: Social: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention: Social | 22.50 [19.00 to 30.00] | 27.00 [23.00 to 36.00]
  Follow-up: Social Composite Score: number analyzed (Participants) | 14 | 15
  Follow-up: Social Composite Score | 22.50 [18.00 to 25.00] | 28.00 [26.00 to 36.00]
  Visit 1 - First Intervention: Speech | 4.00 [2.00 to 8.00] | 7.00 [2.00 to 10.00]
  Visit 2 - First Intervention: Speech | 3.00 [1.00 to 9.00] | 5.00 [2.00 to 11.00]
  Visit 3 - First Intervention: Speech | 5.00 [1.00 to 6.00] | 8.00 [2.00 to 11.00]
  Visit 4 - First Intervention: Speech | 5.50 [3.00 to 8.50] | 5.00 [2.00 to 10.50]
  Visit 5 - First Intervention: Speech | 6.50 [3.00 to 7.50] | 8.00 [2.00 to 11.50]
  Visit 6 - Second Intervention: Speech | 4.00 [1.00 to 6.00] | 8.50 [2.00 to 11.50]
  Visit 7 - Second Intervention: Speech: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention: Speech | 4.00 [2.00 to 5.00] | 7.00 [4.00 to 12.00]
  Visit 8 - Second Intervention: Speech: number analyzed (Participants) | 15 | 14
  Visit 8 - Second Intervention: Speech | 5.00 [1.00 to 7.00] | 6.50 [2.00 to 9.00]
  Visit 9 - Second Intervention: Speech | 5.00 [2.00 to 8.50] | 5.00 [2.00 to 10.00]
  Visit 10 - Second Intervention: Speech: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention: Speech | 5.00 [3.00 to 7.00] | 7.25 [2.50 to 11.00]
  Follow-up: Speech Composite Score: number analyzed (Participants) | 14 | 14
  Follow-up: Speech Composite Score | 6.00 [2.00 to 9.50] | 6.00 [2.00 to 10.50]
  Visit 1 - First Intervention: Symbolic | 9.50 [6.50 to 12.50] | 14.00 [12.50 to 19.50]
  Visit 2 - First Intervention: Symbolic | 10.50 [6.00 to 13.50] | 14.50 [11.00 to 17.00]
  Visit 3 - First Intervention: Symbolic | 10.50 [4.00 to 13.00] | 15.00 [10.00 to 21.00]
  Visit 4 - First Intervention: Symbolic | 12.00 [5.50 to 13.50] | 14.00 [11.50 to 22.00]
  Visit 5 - First Intervention: Symbolic | 11.50 [7.00 to 17.50] | 16.50 [11.50 to 23.00]
  Visit 6 - Second Intervention: Symbolic | 13.00 [6.50 to 15.00] | 18.50 [12.00 to 23.00]
  Visit 7 - Second Intervention: Symbolic: number analyzed (Participants) | 14 | 15
  Visit 7 - Second Intervention: Symbolic | 10.25 [6.00 to 13.00] | 17.00 [10.00 to 22.00]
  Visit 8 - Second Intervention: Symbolic: number analyzed (Participants) | 15 | 14
  Visit 8 - Second Intervention: Symbolic | 11.50 [6.50 to 15.50] | 17.00 [9.00 to 20.50]
  Visit 9 - Second Intervention: Symbolic | 11.50 [9.00 to 18.50] | 18.00 [12.50 to 20.50]
  Visit 10 - Second Intervention: Symbolic: number analyzed (Participants) | 14 | 14
  Visit 10 - Second Intervention: Symbolic | 13.75 [8.00 to 17.00] | 17.00 [11.00 to 19.00]
  Follow-up: Symbolic Composite Score: number analyzed (Participants) | 14 | 14
  Follow-up: Symbolic Composite Score | 14.25 [9.00 to 16.00] | 18.00 [13.50 to 19.00]

16. Secondary Outcome: Aberrant Behavior Checklist - Community Edition (ABC-C)
Description: The ABC-C is a global behavior checklist implemented for the measurement of drug and other treatment effects in populations with intellectual disability. Behavior based on 58 items that describe various behavioral problems.
  Each item is rated on the parents perceived severity of the behavior. The answer options for each item are:
  0 = Not a problem
  1. = Problem but slight in degree
  2. = Moderately serious problem
  3. = Severe in degree
  The measure is broken down into the following subscales with individual ranges as follows:
  Subscale I (Irritability): 15 items, score range = 0-45 Subscale II (Lethargy): 16 items, score range = 0-48 Subscale III (Stereotypy): 7 items, score range = 0-21 Subscale IV (Hyperactivity): 16 items, score range = 0-48 Subscale V (Inappropriate Speech) was not included in the breakdown because it was not applicable (no participants in the study had verbal language).
Time Frame: Every 5 weeks during each of the two 20-week treatment periods, and once 4 weeks after final treatment ends
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  Visit 1 - First Intervention: Subscale I | 9.00 [6.00 to 22.00] | 6.00 [3.00 to 12.00]
  Visit 3 - First Intervention: Subscale I | 9.00 [2.00 to 15.00] | 4.00 [0.00 to 7.00]
  Visit 5 - First Intervention: Subscale I | 7.00 [0.00 to 16.00] | 2.00 [0.00 to 6.00]
  Visit 6 - Second Intervention: Subscale I | 7.00 [3.00 to 13.00] | 4.00 [0.00 to 10.00]
  Visit 8 - Second Intervention: Subscale I | 4.00 [1.00 to 17.00] | 3.00 [0.00 to 10.00]
  Visit 10 - Second Intervention: Subscale I: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Subscale I | 5.00 [2.00 to 14.00] | 5.00 [0.00 to 8.00]
  Follow-up: Subscale I (Irritability): number analyzed (Participants) | 15 | 13
  Follow-up: Subscale I (Irritability) | 3.00 [0.00 to 9.00] | 2.00 [0.00 to 7.00]
  Visit 1 - First Intervention: Subscale II | 13.00 [5.00 to 19.00] | 8.00 [4.00 to 10.00]
  Visit 3 - First Intervention: Subscale II | 11.00 [3.00 to 17.00] | 7.00 [3.00 to 8.00]
  Visit 5 - First Intervention: Subscale II | 9.00 [5.00 to 12.00] | 6.00 [4.00 to 10.00]
  Visit 6 - Second Intervention: Subscale II | 11.00 [5.00 to 16.00] | 5.00 [2.00 to 9.00]
  Visit 8 - Second Intervention: Subscale II | 8.00 [4.00 to 11.00] | 5.00 [2.00 to 9.00]
  Visit 10 - Second Intervention: Subscale II: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Subscale II | 6.00 [4.00 to 9.00] | 4.00 [2.00 to 6.00]
  Follow-up: Subscale II (Lethargy): number analyzed (Participants) | 15 | 13
  Follow-up: Subscale II (Lethargy) | 6.00 [2.00 to 11.00] | 5.00 [2.00 to 8.00]
  Visit 1 - First Intervention: Subscale III | 13.00 [10.00 to 16.00] | 12.00 [9.00 to 14.00]
  Visit 3 - First Intervention: Subscale III | 10.00 [8.00 to 15.00] | 10.00 [8.00 to 13.00]
  Visit 5 - First Intervention: Subscale III | 11.00 [9.00 to 16.00] | 9.00 [7.00 to 12.00]
  Visit 6 - Second Intervention: Subscale III | 11.00 [7.00 to 16.00] | 11.00 [9.00 to 12.00]
  Visit 8 - Second Intervention: Subscale III | 10.00 [7.00 to 15.00] | 9.00 [7.00 to 11.00]
  Visit 10 - Second Intervention: Subscale III | 8.00 [6.00 to 12.00] | 9.00 [7.00 to 12.00]
  Follow-up: Subscale III (Stereotypy) | 8.00 [6.00 to 11.00] | 9.00 [7.00 to 12.00]
  Visit 1 - First Intervention: Subscale IV | 13.00 [8.00 to 22.00] | 8.00 [6.00 to 14.00]
  Visit 3 - First Intervention: Subscale IV | 12.00 [7.00 to 15.00] | 8.00 [3.00 to 13.00]
  Visit 5 - First Intervention: Subscale IV | 11.00 [8.00 to 26.00] | 6.00 [3.00 to 6.00]
  Visit 6 - Second Intervention: Subscale IV | 11.00 [7.00 to 22.00] | 7.00 [2.00 to 17.00]
  Visit 8 - Second Intervention: Subscale IV | 7.00 [5.00 to 16.00] | 4.00 [0.00 to 11.00]
  Visit 10 - Second Intervention: Subscale IV: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Subscale IV | 10.00 [4.00 to 20.00] | 5.00 [2.00 to 10.00]
  Follow-up: Subscale IV (Hyperactivity): number analyzed (Participants) | 15 | 13
  Follow-up: Subscale IV (Hyperactivity) | 9.00 [3.00 to 17.00] | 5.00 [1.00 to 9.00]

17. Secondary Outcome: Quantitative Measures of Respiration: Apnea Index
Description: Respiratory data was collected using non-invasive respiratory inductance plethysmography from a BioCapture® recording device. BioCapture® is a child-friendly measurement device that can record from 1 to 12 physiological signal transducers in a time-locked manner. It can be configured with the pediatric chest and abdominal plethysmography bands and the 3 lead ECG signals we plan to use for monitoring cardiac safety throughout the study. Each transducer is placed on the patient independently to provide a customized fit that yields the highest signal quality for each patient irrespective of body shape and proportion. The transducer signals captured by the BioCapture® are transmitted wirelessly to a laptop computer where all signals are displayed in real-time.
  The apnea index is given as apneas/hour. Data on apneas greater than or equal to 10 seconds are displayed below. The higher the frequency of apnea, the more severe the breathing abnormality.
Time Frame: Every 10 weeks during each of the two 20-week treatment periods
Population: In some cases, the number of participants analyzed is less than 15 for each group due to inability to complete testing session.
  One participant from the "rhIGF-1 First, Then Placebo" group was removed from the study prior to Visit 10, so there is only data for 14 participants included at that time point.
Measure: Median (Inter-Quartile Range); unit: Apneas/Hour
Arm/Group | Placebo First, Then rhIGF-1 | rhIGF-1 First, Then Placebo
Number analyzed (Participants) | 15 | 15
Apneas/Hour
  Visit 1 - First Intervention: Apnea Index: number analyzed (Participants) | 15 | 14
  Visit 1 - First Intervention: Apnea Index | 7.58 [1.58 to 10.33] | 4.05 [2.07 to 7.91]
  Visit 3 - First Intervention: Apnea Index: number analyzed (Participants) | 15 | 14
  Visit 3 - First Intervention: Apnea Index | 4.80 [0.38 to 9.20] | 3.48 [2.00 to 4.19]
  Visit 5 - First Intervention: Apnea Index: number analyzed (Participants) | 15 | 14
  Visit 5 - First Intervention: Apnea Index | 6.93 [3.06 to 9.07] | 3.07 [0.40 to 5.11]
  Visit 6 - Second Intervention: Apnea Index: number analyzed (Participants) | 15 | 14
  Visit 6 - Second Intervention: Apnea Index | 7.90 [4.30 to 17.60] | 3.62 [2.20 to 11.82]
  Visit 8 - Second Intervention: Apnea Index: number analyzed (Participants) | 15 | 14
  Visit 8 - Second Intervention: Apnea Index | 7.28 [2.80 to 12.53] | 5.55 [1.24 to 12.81]
  Visit 10 - Second Intervention: Apnea Index: number analyzed (Participants) | 15 | 14
  Visit 10 - Second Intervention: Apnea Index | 8.91 [4.13 to 14.34] | 5.56 [1.57 to 13.47]

ADVERSE EVENTS:
Time Frame: 80 weeks (from screening visit to 12-week follow up phone call).
Groups:
- Placebo: This group includes subjects who had a reported Adverse Event (AE) while they were receiving placebo treatment.
- rhIGF-1: This group includes subjects who had a reported Adverse Event (AE) while they were receiving rhIGF-1 treatment.
- Off Treatment: This group includes subjects who had a reported Adverse Event (AE) while they were not receiving any treatment. This includes the period between Screening and Baseline, the 20-week washout period between study arms, and the 12-week follow up period after study completion.
Arm/Group | Placebo | rhIGF-1 | Off Treatment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 4/30 | 2/30
Other Adverse Events (participants affected / at risk) | 16/30 | 20/30 | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=30) | rhIGF-1 (N=30) | Off Treatment (N=30)
Colitis (Gastrointestinal disorders) | 0/15 (0) | 1/15 (1) | 0 (0)
Seizure (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | rhIGF-1 (N=30) | Off Treatment (N=30)
Abnormal ECG - Prolonged QT (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Adenoidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Advanced Bone Age (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Otitis Media (Ear and labyrinth disorders) | 2 (2) | 4 (4) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Precocious Puberty (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Seizures (General disorders) | 3 (4) | 1 (1) | 2 (2)
Seizure and Fever (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Seizure and vomiting (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Vomiting and Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Elevated Alkaline Phosphatase (General disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive Cough and Vomiting (General disorders) | 1 (1) | 0 (0) | 0 (0)
Car Accident (General disorders) | 0 (0) | 0 (0) | 1 (1) — Participant was in car accident on way to study visit. No injuries sustained.
Extrapyramidal Disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrostomy Tube Replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hand, Foot, and Mouth Disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Minor Head Injury (General disorders) | 0 (0) | 1 (1) | 0 (0)
Other Cardiac Disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Personality Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin (Eye) Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar Hypertrophy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Unequal limb length (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No